CLINICAL TRIAL: NCT06808360
Title: Supportive and Dignified Maternity Care (SDMC) - Development and Feasibility Assessment of an Intervention Package for Public Health Systems
Brief Title: Supportive and Dignified Maternity Care in Public Health Facilities
Acronym: SDMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Karachi (Other)
Responsible Party: Principal Investigator, Waqas Hameed, Senior Instructor, Aga Khan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Aku2020
Record Dates: First submitted 2025-01-28; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2021-04

CONDITIONS: Behavior, Health
MeSH Terms: conditions — Health Behavior | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: SDMC is a theory-driven, inclusive service-delivery package developed using the principles of the human-centered design approach. The model will focus on capacity-building for maternity teams and improving governance and accountability mechanisms within public health facilities. This ensures that all women are treated with compassion and dignity, while also addressing their diverse needs, including disabilities and common mental health conditions. A unique feature of the intervention package is the integration of psychosocial support into routine maternity care, with a principal aim of addressing the psychological needs of birthing women and their companions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive and Dignified Maternity Care (SDMC) (Experimental): Maternity staff at six health facilities will be exposed to the intervention package. The intervention will be evaluated using a pre-post comparison design.
  Interventions: Behavioral: Supportive and Dignified Maternity Care

INTERVENTIONS:
Behavioral: Supportive and Dignified Maternity Care — SDMC is a theory-driven, inclusive service-delivery package which will be developed using the principles of the human-centred design approach. The model will include capacity-building of maternity teams, and the improvement of governance and accountability mechanisms within public health facilities to ensure that all women are treated with compassion and dignity, while also catering for their diverse needs, including disabilities and common mental health conditions. The integration of psychosocial support in routine maternity care will be a unique feature of the intervention package, a principal aim of which is to address the psychological needs of birthing women and their companions.

SUMMARY:
Brief Summary Poor psychosocial support and demeaning care during childbirth in health facilities are common worldwide, particularly in low- and middle-income countries. Despite a policy directive from the World Health Organization (WHO), there is no operational model that effectively demonstrates the incorporation of these guidelines into routine facility-based maternity services. Recent evidence from Pakistan highlights a high rate of reported disrespect and abuse during childbirth, with several health system factors contributing to this compromised care.

This early-phase research aims to develop, implement, and test the feasibility of a Supportive and Dignified Maternity Care (SDMC) service-delivery model. Based on WHO's guiding principles and framework, the model promotes respectful and supportive intrapartum care in public health facilities. The components of the SDMC model include:

Participatory and co-created service-delivery intervention;

Capacity-building of maternity teams (clinical and support staff) through a partnership approach;

Collaborative Care Model;

Patient orientation in the processes of care and their SDMC rights;

Information system (e.g., complaints register);

Accountability mechanisms (e.g., exit interviews); and

Embedding performance reviews.

Using a mixed-method design and extensive data collection before, during, and after the implementation of the intervention, we will assess the coverage of the intervention and its fidelity-the extent to which SDMC guidelines are being adhered to. Challenges faced, changes in maternity teams' understanding and attitudes, and improvements in women's maternity experiences and psychosocial well-being will also inform the success of the intervention.

Evidence from this research will guide further refinements to the SDMC model package. It will provide insights into behavior change among maternity staff and birthing women, as well as estimate the potential effect size to design a larger evaluation and scalability research in diverse health system contexts.

DETAILED DESCRIPTION:
Background:

Respectful and dignified healthcare is a fundamental right for every woman. However, in health facilities, particularly in low- and middle-income countries, women's experiences of maternity care are often characterized by discrimination, poor psychosocial support, and patronizing attitudes from service providers. Such distressing encounters during obstetric care are likely to have adverse effects on both women and newborns. Women with disabilities and mental health needs are especially vulnerable to poor care and the suffering it causes.

Goal and Objectives:

To support inclusive Supportive and Dignified Maternity Care (SDMC) within health systems, particularly from the perspective of:

1. The capacity of service providers, and
2. Accountability and governance.

The specific objectives are to:

ASSESS: Health system challenges and opportunities for inclusive, supportive, and dignified intrapartum care.

DESIGN: A service-delivery model through a participatory, consensus-driven process.

TEST: The feasibility of the model for content and operationalization in health facilities.

Intervention:

The components of the SDMC model include:

Co-created implementation strategy;

Capacity-building of maternity teams (clinical and support staff);

Collaborative care;

Staff and patient feedback; and

Accountability and governance (performance review).

Methods:

The project will span a period of twenty-four months. Using a mixed-method design, data will be collected at different time intervals to assess the feasibility of the intervention. Challenges faced during implementation, changes in maternity teams' understanding and attitudes, and improvements in women's maternity experiences will also inform the success of the intervention.

Expected Outcomes:

A handbook for capacity-building of health facility staff to provide inclusive and dignified maternity care.

An adapted mhGAP manual for labor room staff to provide birthing women with psychosocial support.

An implementation strategy for embedding inclusive SDMC principles within public health systems.

Contextually adapted measurement tools for inclusive, supportive, and dignified care.

ELIGIBILITY:
Postnatal Women

Inclusion Criteria:

Delivered in a study health facility during the data collection period.

Provided informed consent.

Exclusion Criteria:

Reside outside the demarcated catchment area.

Health Facility Staff

Inclusion Criteria:

Employed at the study health facility.

Provided informed consent.

Exclusion Criteria:

Recently appointed to the health facility (less than 6 months).

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 314 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Mean score of women's experiences of supportive and dignified maternity care | Women will be interviewed at baseline. It will follow a six month intervention period. At the end of intervention endline survey will be conducted somewhere Sep - Dec 2021.
  The Women's experiences of SDMC will be assessed using a Mistreatment standard tool that will be adapted in the Pakistani context. The score range will be 0-100 where a higher score will indicate higher level of mistreatment whereas lower score will reflect better care.

SECONDARY OUTCOMES:
Perception of service providers about feasibility of SDMC intervention | Endline assessment that will be done at the end of a six month intervention period. The assessment will be done in September-November 2021.
  Service providers will be qualitative enquired about their experiences of training and how feasible they found to implement the intervention. They will be asked about challenges and suggestions for improvements

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Iqbal Avan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Thatta Project Office, Thatta, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
This is under discussion.